CLINICAL TRIAL: NCT03955653
Title: Fluoroscopic-Guided Micropuncture Technique for Common Femoral Artery Access: Comparisons of Oblique vs. Antero-Posterior Projections for Femoral Artery Access
Brief Title: Fluoroscopic-Guided Micropuncture Technique for Common Femoral Artery Access
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Massoud Leesar, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRB-300001879
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-05

CONDITIONS: Catheter Related Complication

STUDY DESIGN:
Intervention Model Description: Patients will be randomized equally to the right anterior oblique view using fluoroscopy and the access to the femoral artery will be compared to that in the anterior-posterior projection
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAO projection (Active Comparator): Patients will be randomized to right anterior oblique (RAO) projection by fluoroscopy for the access to the femoral artery
  Interventions: Procedure: Femoral artey access
- AP projection (Active Comparator): Patients will be randomized to anterior-posterior projection by fluoroscopy for the access to the femoral artery
  Interventions: Procedure: Femoral artey access

INTERVENTIONS:
Procedure: Femoral artey access — We will study the access to the femoral artery for cardiac catheterization or percutaneous coronary intervention

SUMMARY:
The main objective of this proposed study is to examine if oblique projection (20- degrees right anterior oblique (RAO) for right femoral artery access or 20-degree left anterior oblique (LAO) for left femoral artery access) is superior to anterior projection (AP) for femoral artery access in zone 2-4 and thereby resulting in lower risk of access related complications.

DETAILED DESCRIPTION:
The investigators plan to randomize 200 subjects who present for coronary angiography, bypass graph angiography or left heart catheterization via the femoral approach. The investigators will randomly assign them to either oblique projection (20-degree RAO for right femoral artery) or 20-degree LAO (for left femoral artery) versus AP for femoral arterial access in a 1:1 fashion. A trained cardiologist will review the femoral artery angiogram. The investigators will use the scoring system used for the femoral artery access site, as previously reported (10). These predefined locations are as follows: zone 1 denotes femoral artery above the femoral head; zone 2, femoral artery from the superior border of femoral head to the center of the femoral head; zone 3, femoral artery in the center of the femoral head; zone 4, femoral artery from the center of femoral head to the inferior border of the femoral head; and zone 5, femoral artery below the inferior boarder of the femoral head.

The invesigators will use micropuncture access kit for femoral artery access. Micropuncture needle will be advanced to the center of the femoral head and common femoral artery will be punctured guided by fluoroscopy. Those assigned to oblique projection will have fluoroscopic-guided femoral access in RAO 20 degree for right femoral artery and LAO 20 degree for left femoral artery, while those assigned to AP will have femoral artery access in AP 0 degree. For both groups, the investigators will also obtain the other view as a reference to compare results (i.e., in the oblique group, we will save AP and vice versa). If the tip of the micropuncture needle were located in the femoral artery corresponding to the center (zone 3) or bottom third (zone 4) of the femoral head in the 20-degree RAO, 20-degree LAO position or zero-degree AP position, the micropuncture dilator will be advanced into the femoral artery, 0.018" guide wire will be exchanged with a 0.035" guide wire, and a sheath will be placed in the femoral artery, and the femoral angiography will be performed in the 20-degree RAO or 20-degree LAO projection for right and left femoral artery, respectively.

The investigators will also collect data on demographic characteristics including age, race, gender, as well as cardiovascular risk factors such as history of diabetes, hypertension, dyslipidemia, peripheral arterial disease, prior CAD, prior CVA, smoking history, family history of CAD, eGFR. We will also obtain data on medication history to review if they are on antiplatelet or anticoagulants. Those with ipsilateral access within the past 90 days will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing cardiac catheterization or PCI

Exclusion Criteria:

* Peripheral vascular disease
* Renal failure, Creatinine >2.5 mg/dL
* Hemodynamic instability, acute myocardial infarction
* Heart failure with EF<25%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The percentage of access to the central portion of the femoral artery (Zone III) | the procedure
  We will assess the access to the center of the femoral artery after insertion of the sheath for heart catheterization or PCI
The success rate of access to the Zone III | the procedure
  We will define the access to the zone III with angiography

SECONDARY OUTCOMES:
The rate of access site complications | the procedure
  Hematoma, bleeding complication, femoral artery dissection, pseudoaneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Massoud A Leesar, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leesar MA, Waheed S, Al Solaiman F, Chatterjee A, Daya HA, Hage FG, Brott BC. Randomized trial of an oblique versus standard fluoroscopic-guided micropuncture technique for femoral arterial access: The Micropuncture-CFA trial. Cardiovasc Revasc Med. 2023 Dec;57:43-50. doi: 10.1016/j.carrev.2023.06.029. Epub 2023 Jun 28. PMID 37414613